CLINICAL TRIAL: NCT04701996
Title: Transmission Dynamics of COVID-19 in a Rural Setting of the Democratic Republic of the Congo
Acronym: DynaCovid
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Centre de Recherche en Santé de Kimpese (Unknown); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Other Study IDs: B3002020000141
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: serological test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort: sero-surveillance will start in a cohort of 800 adults (18-50y). In case of an established outbreak, this sample will be extended to 400 children (0-17y) and 400 elderly (50+y).
  Interventions: Biological: serological surveillance

INTERVENTIONS:
Biological: serological surveillance — serological surveillance, detection of antibodies (Total Ig and IgM) developed against SARS-CoV-2 in a population living in a rural area (Kimpese, DRC)

SUMMARY:
A fixed cohort of adults in rural Kimpese will be followed up every two months since they are assumed to be at above average risk of contracting COVID-19. Every two months these individuals will be interviewed with a focus on COVID-19 related symptoms and possible exposure to the disease and have their temperature recorded.

A social mixing survey will also be carried out to assess human contact behaviour. The data generated will help inform mathematical modelling that can predict which proportion of the population per age group is likely to get infected once COVID-19 is introduced in this rural population, and the epidemic size if no intervention, as well as when targeted interventions are introduced. During the outbreak, physical distancing measures could be implemented. The monitoring of social contacts, again using a social-mixing survey, will contribute to the understanding of the impact of such measures in a rural context on transmission of SARS-CoV-2. The results from the seroprevalence over time, will be used to refine and validate the predictions from the modelling results, (re)calibrate the model where needed, and test hypotheses on transmission-dynamics of COVID-19.

In case of an established epidemic of Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in the Health Zone of Kimpese, the sero-surveillance will be extended from an assumed high risk cohort to a representative sample of the overall population. Moreover, support to the COVID-19 control measures will be provided by the study team. The national guidelines recommend household transmission investigation for the first 100 confirmed laboratory cases. During the household visit, information on symptoms and one serum sample will be requested of all household members of the index case. If household members are present with symptoms and fever, the COVID-19 outbreak team of Kimpese will provide diagnostic testing and medical care.

DETAILED DESCRIPTION:
The sero-surveillance will start in a cohort of 800 adults (18-50y). In case of an established outbreak, this sample will be extended to 800 pre-school children (0-5y), 800 schoolchildren (6-17y) and elderly (50+y). Human interactions will be quantified for the rural context of Kimpese in four age categories, pre-school children (0-5y), schoolchildren (6-17y), adults (18-50y) and elderly (50+). A sample of 300 persons in each age group will be selected.

The study site will be the Health Demographic Surveillance System (HDSS) in the health district of Kimpese, Kongo-Central province, DRC, managed Centre de Recherche en Santé de Kimpese (CRSK). Each village, household and household member is listed in the HDSS database, each household has been geo-referenced. The HDSS has enrolled a cohort of 60 000 inhabitants in 11 rural health areas of the district. CRSK is the partner involved in the study and from the core database the cohort population for the study will be selected using two stage sampling. In stage one 20 villages will be randomly selected from the HDSS database using population size as sampling weight. In stage two a random sample of 40 eligible individuals will be drawn in each of the selected villages.

In the cohort, a blood sample will be collected for serology (sero-surveillance). When an individual presents seroconversion, the household attack rate will be explored. Information on symptoms and one serum sample of each household member, irrespective of age, will be requested during the next follow-up visit. Any study subject reporting symptoms or presenting with a fever, will be referred to the Institut Médical Evangélique (IME) hospital for appropriate medical care.

A social mixing survey will be carried out to assess human contact behaviour, in an extended cohort involving four age groups (0-5 years; 6-17 years; 18-50 years; >50 years old), sampled from the overall population in rural Kimpese.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for the sero-survey, study participants must meet the following criteria:

* Resident of the Kimpese HDSS demographic surveillance area
* Adults 18-50 years old
* When SARS-CoV-2 transmission is confirmed, all ages will be eligible to participate
* Willing and able to provide written informed consent

In order to be eligible for the social-mixing survey, study participants must meet the following criteria:

* Resident of the Kimpese HDSS demographic surveillance area
* Willing and able to provide written informed consent

Exclusion Criteria:

* refusal to participation

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study site will be the Health Demographic Surveillance System (HDSS) in the health district of Kimpese, Kongo-Central province, DRC, managed by Centre de Recherche en Santé de Kimpese (CRSK). Each village, household and household member is listed in the HDSS database, each household has been geo-referenced. The HDSS has enrolled a cohort of 60 000 inhabitants in 11 rural health areas of the district. Up to now, this area has not declared any COVID-19 cases. The IME hospital of Kimpese has been designated for the hospitalisation and medical care of COVID-19 suspect and confirmed cases and the outbreak response team has been established
Sampling Method: Probability Sample
Enrollment: 1709 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To predict and monitor the transmission of SARS-CoV-2 in a rural Sub Saharan setting. | 1 year
  qualitative and quantitative monitoring of antibody response against SARS-CoV-2. Wantai SARS CoV-2 (Ig + IgM) is used for the detection of total Ig and IgM antibodies against SARS-CoV-2. This assay allows for qualitative (antibodies present or absent) and quantitative detection of antibodies. The amount of colour intensity is measured and is proportional to the amount of antibody captured inside the wells, and to the sample respectively (quantitative result)
To inform intervention strategies targeted at limiting the spread of COVID-19 in a rural Sub Saharan setting. | 1 year
  To combine all information to inform dynamic transmission model that can simulate the spread of SARS-CoV-2 and the effect of intervention strategies to inform public health policy.

SECONDARY OUTCOMES:
To create social contact matrices that can be used to parameterise dynamic transmission models. | 1 year
  To assess the change in social mixing patterns following the introduction of COVID-19 related physical distancing measures

OTHER OUTCOMES:
To identify risk factors of SARS-CoV-2 infection in a rural Sub Saharan setting | 1 year
  The combination of sero-surveillance and social mixing results will provide elements for mathematical modelling that can predict which proportion of the population per age group is likely to get infected once COVID-19 is introduced in this rural population

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Inocencio da Luz, PhD, Principal Investigator — Insitute of Tropical Medicine
Locations (1):
- Centre de Recherche en Santé de Kimpese, Kimpese, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided